CLINICAL TRIAL: NCT06839027
Title: Arterial to Central Venous co2 Gap in Relation to Outcome After Cardiopulmonary Bypass
Brief Title: Arterial to Central co2gap in Relation to Outcome After Cardiopulmonary Bypass
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marina emad fawzi hanna, doctor holding masters degree in anathesia and icu, Ain Shams University
Other Study IDs: FMASU MD305/2024
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-04

CONDITIONS: Patient Undergoing CABG Surgery; Ischemic Heart Disease Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- survival group and mortality group: patients will be categorized into two groups (mortality VS survival group)

SUMMARY:
This trial aims to study the performance of CO2 gap, lactate level, and central venous oxygen saturation in predicting major postoperative complications after cardiac surgery with cardiopulmonary bypass

DETAILED DESCRIPTION:
Complications after cardiac surgery (e.g., acute respiratory failure, circulatory failure, acute kidney injury, neurological failure, etc.) are associated with high morbidity and mortality .

One crucial cause is the mismatch of oxygen delivery and consumption after the surgery, which is often the result of a decrease in cardiac output and/or an increase in oxygen demand due to stress . The imbalance of oxygen delivery and consumption leads to tissue hypoxia. Organ injury and dysfunction can occur if tissue hypoxia is not corrected. Timely identification and management of tissue hypoxia are essential to prevent the development of organ dysfunction and postoperative complications. Several biomarkers of hypoxia have been proposed to identify tissue hypoxia.

Markers of adequate tissue perfusion (lactate, ScVO2, and CO2 gap) have their limitations. Hyperlactatemia does not always reflect tissue dysoxia or anaerobic metabolism and can be aspecific (Schultz et al., 2006). Central venous oxygen saturation (ScVO2), used as a marker of dysoxia, can be normal despite microcirculatory impairment (Habicher et al., 2015). CO2 gaps can be used as a surrogate for the adequacy of cardiac output (CO) and as a marker for tissue perfusion and are therefore a potential target for resuscitation.

Current examinations are not satisfactory enough to answer the question of adequacy between oxygen supply and demand. Urine output, at its best, reflects the function of one organ only. The mixed venous oxygen saturation (SvO2) and the central venous oxygen saturation (ScvO2) reflect the oxygen exertion rate. However, they are often in a normal range or even in a supra-normal level in septic shock despite the presence of tissue anaerobic metabolism, partly due to microcirculatory shunting or the inability of the tissues to use oxygen (i.e., cytopathic hypoxia), or both . CO2-derived parameters overcome many of the limitations of the previous indices in indicating anaerobic tissue metabolism ,one can briefly interpret the concept as follows: the venous-arterial difference in CO2 partial pressure (Pv-aCO2 or PCO2 gap) is a useful index of the adequacy of cardiac output (CO) for the global metabolic conditions. In other words, a decrease in CO results in an increased PCO2 gap and vice versa. It can be measured as a venoarterial difference in PCO2 (PvCO2 - PaCO2).

CPB is a form of extracorporeal circulation whose function is to maintain circulation and respiratory support along with temperature management to facilitate operation on the heart and great vessels.

Components of the CPB machine include pumps, tubing, gas (oxygenator), and heat exchange units. Modern CPB machines are also equipped with monitoring systems that continuously monitor line or circuit pressure, temperature, and blood parameters (oxygen saturation, blood gases, hemoglobin [Hgb], potassium), as well as safety features such as air bubbles and fluid level detection systems and a blood filter in the arterial line .

CPB mechanically circulates and oxygenates blood for the body while bypassing the heart and lungs. The surgeon places a cannula in the right atrium, vena cava, or femoral vein to withdraw blood. Venous blood which is removed from the body by the venous cannula is filtered, cooled or warmed, oxygenated, and then returned to the body. The arterial cannula used to return oxygenated blood is usually inserted in the ascending aorta, but it may be inserted in the femoral artery. During the procedure, hypothermia may be maintained; body temperature is usually kept at 28 °C to 32 °C. The blood is cooled during CPB and returned to the body.

The PCO2 gap is the difference between the partial pressure of CO2 in venous blood (PvCO2) and arterial blood (PaCO2). PCO2 gap is considered to be a marker of the relationship between cardiac output (CO) to global metabolic demand, a marker of adequacy of venous blood flow to eliminate CO2 produced by peripheral tissues. Considering physiology, CO2 is the end product of aerobic metabolism and therefore venous CO2 content thus, PCO2 reflects the global tissue blood flow relative to metabolic demand. Under steady-state conditions, the PCO2 gap is determined by several factors: difference in veno-arterial CO2 content, CO2 dissociation curve (which expresses the relationship between CO2 pressure and CO2 content), CO, and alveolar ventilation. It has been shown that out of all these factors, a fall in CO has the maximum influence on the CO2 gap .

ELIGIBILITY:
Inclusion Criteria:

* • Patients undergoing elective cardiac surgery (Cardiopulmonary Bypass Grafting), with a maximum time on cardiopulmonary bypass of 120 minutes, will be screened for study eligibility.

  * The inclusion criteria are:

    1. Age ≥ 18.
    2. Receive elective cardiac surgery (CABG) involving CPB with maximum time on CPB 120 mins.
    3. Admitted to ICU after the surgery.
    4. With an arterial line and a central venous catheter in place.

       Exclusion Criteria:

    <!-- -->

    1. Unwilling to provide consent.
    2. Acute or chronic kidney disease before surgery
    3. Acute or chronic hepatic insufficiency before surgery.
    4. Malpositioning of the central venous catheter
    5. Pregnant.
    6. Patients with respiratory disorders such as COPD.
    7. Patients with a BMI more than or equal to 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing single cardiac surgery on bypass and post-operative in ICU for 7 days.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-05-02 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
7 days mortality | 7 days
  patients will be followed up for 7 days post operative

SECONDARY OUTCOMES:
1) Duration of mechanical ventilation. 2) Length of ICU stays. 3) Acute kidney injury (AKI). 4) Myocardial infarction. 5) Circulatory shock for any cause, | 7 days
  1. Duration of mechanical ventilation.
  2. Length of ICU stays.
  3. Acute kidney injury (AKI).
  4. Myocardial infarction.
  5. Circulatory shock for any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt